CLINICAL TRIAL: NCT03373513
Title: Robotic-assisted Hysterectomy: Single- vs. Multi-port Laparoscopic Access
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: hospital never sterted on single site laparoscopy
Sponsor: Herning Hospital (Other)
Responsible Party: Principal Investigator, Finn Lauszus, Research Specialist, Senoir Consultant, Assistant Professor, Herning Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-SSH
Record Dates: First submitted 2017-12-07; First posted 2017-12-14 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Activity, Motor; Pain; Wound
Keywords: Return-to-work, Visual analogue pain score, Cosmesis
MeSH Terms: conditions — Motor Activity; Pain; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Women are randomized to either robotic single site or multi port lapsoscopic hystrectomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic single-site hysterectomy (Active Comparator): Robotic single-site hysterectomy is performed in this arm
  Interventions: Procedure: Robotic single-site Hysterectomy
- Multiport Laparoscopy (Active Comparator): Multiport Laparoscopic hysterectomy is performed in this other arm
  Interventions: Procedure: Laparoscopic hysterectomy

INTERVENTIONS:
Procedure: Robotic single-site Hysterectomy — Robotic assisted Periumbilical single incision hysterectomy
  Arms: Robotic single-site hysterectomy
Procedure: Laparoscopic hysterectomy — Multiport laparoscopic hysterectomy
  Arms: Multiport Laparoscopy

SUMMARY:
robotic single site surgery (R-SSH) is a novel technique, which may be superior to conventional multiport hysterectomy in select patients regarding cosmesis and postoperative pain. We, perform a randomized trial to compare R-SSH with multiport laparoscopic hysterectomy with regard to the postoperative rehabilitation, cosmesis, the operational cost, and the perioperative morbidity.

DETAILED DESCRIPTION:
The study is scheduled to start February 2018 and compares robotic single-site hysterectomy to conventional multiport hysterectomy. Procedures are performed by an experienced two-surgeon team. Patients are randomized to either conventional multiport hysterectomy (N=62) or R-SSH (N=62). Eligibility criteria are the same as for study 1. Patient's satisfaction with body image and cosmesis is assessed at different time points pre- and postoperatively by means of validated cosmesis scales and Body Image Questionnaire. Postoperative pain and analgesia use will be registered as well as secondary outcome parameters as described above. A follow-up at 1, 3 and 6 month include evaluation of the scar and registration of port-site hernias and vaginal dehiscence or other complications. Interviews and diaries will include time of return to home and work, daily activities including sexuality The R-SSH is performed using da Vinci, Xi robotic system. One single port, diameter 2 cm is applied. Applying an additional assistant port is defined conversion of procedure The laparoscopy is performed using our standard equipment and 4 trocars, 5 mm each.

Socio-economical consequences of R-SSH versus conventional laparoscopic hysterectomy Study details in preparation

Sample size calculation was based a previous study on fast track hysterectomy, which showed a difference in return to work of 4 days. 62 women in each group is needed with standard deviation ±8 and a power of 80%. To include those not working, we calculated that with an expected visual analog pain score of 0.86 ±0.2 and 62 in each group the sample was sufficient to detect of difference of 0.1 in visual analog pain score with a power of 80%. All calculation are based on two-sided testing with alpha of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* hysterectomy on benign indication,
* American Society of Anesthetists group 1 or 2,
* BMI less than 35 kg/m2
* uterine size less than 300 g estimated by ultrasound, using Ferraris formula.

Exclusion Criteria:

* adhesions
* prior extensive abdominal surgery
* prior midline incision,
* cutis laxa of abdomen surgery
* endometriosis
* more than 1 cesarean section
* malignant disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women undergoing hysterectomy
Enrollment: 0 (Actual)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Return-to-work | up to six months after operation or until work is resumed, whichever came first
  Time from operation to return work

SECONDARY OUTCOMES:
Pain measured by subjective score | Visual analogue pain score first, second, third, fourth, fifth, and six months after operation
  Visual analogue pain score with a minimum of '0' up to '10' on a 10 cm continious scale

CONTACTS AND LOCATIONS:
Overall Officials: Finn F Lauszus, MD,PhD, Principal Investigator — Gynecology Department, Herning Hospital
Locations (1):
- Gynecology Dept. Herning Hospital, Herning, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
via meeting, posters, abstracts, and publications

REFERENCES:
- [Background] El Hachem L, Andikyan V, Mathews S, Friedman K, Poeran J, Shieh K, Geoghegan M, Gretz HF 3rd. Robotic Single-Site and Conventional Laparoscopic Surgery in Gynecology: Clinical Outcomes and Cost Analysis of a Matched Case-Control Study. J Minim Invasive Gynecol. 2016 Jul-Aug;23(5):760-8. doi: 10.1016/j.jmig.2016.03.005. Epub 2016 Mar 15. PMID 26992935
- [Background] Golkar FC, Ross SB, Sperry S, Vice M, Luberice K, Donn N, Morton C, Hernandez JM, Rosemurgy AS. Patients' perceptions of laparoendoscopic single-site surgery: the cosmetic effect. Am J Surg. 2012 Nov;204(5):751-61. doi: 10.1016/j.amjsurg.2011.07.026. PMID 23140831
- [Background] Sandberg EM, la Chapelle CF, van den Tweel MM, Schoones JW, Jansen FW. Laparoendoscopic single-site surgery versus conventional laparoscopy for hysterectomy: a systematic review and meta-analysis. Arch Gynecol Obstet. 2017 May;295(5):1089-1103. doi: 10.1007/s00404-017-4323-y. Epub 2017 Mar 29. PMID 28357561
- [Background] Yeung PP Jr, Bolden CR, Westreich D, Sobolewski C. Patient preferences of cosmesis for abdominal incisions in gynecologic surgery. J Minim Invasive Gynecol. 2013 Jan-Feb;20(1):79-84. doi: 10.1016/j.jmig.2012.09.008. PMID 23312246
- [Background] Aarts JW, Nieboer TE, Johnson N, Tavender E, Garry R, Mol BW, Kluivers KB. Surgical approach to hysterectomy for benign gynaecological disease. Cochrane Database Syst Rev. 2015 Aug 12;2015(8):CD003677. doi: 10.1002/14651858.CD003677.pub5. PMID 26264829

DOCUMENTS (2):
  • Study Protocol (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT03373513/Prot_001.pdf
  • Informed Consent Form (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT03373513/ICF_000.pdf